CLINICAL TRIAL: NCT03962413
Title: Endoscopic Approaches To The Maxillary Sinus: A Comparative Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa Ibrahem Mohammed, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Approaches To Maxillary Sinus
Record Dates: First submitted 2019-05-19; First posted 2019-05-24 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Maxillary Sinus Surgery
Keywords: Endoscopic Approaches To Maxillary Sinus

STUDY DESIGN:
Intervention Model Description: It is a prospective randomized comparative clinical study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The middle meatal antrostomy approach. (Active Comparator): The middle turbinate will be gently moved medially. Then uncinectomy is the next step which will be performed in numerous ways. Once the natural ostium will be identified, an ostium seeker will be placed through the ostium and then carefully will be pushed posteriorly to widen the ostium.
  Using a through-cutting forceps, the ostium will be enlarged.
  Interventions: Procedure: Endoscopic Approaches To Maxillary Sinus
- The endoscopic prelacrimal recess approach (Active Comparator): A curved incision will be made between the anterior aspect of the IT and the posterior end of the nasal vestibule.the mucoperiosteum will be lifted posteriorly.Bone removal will be achieved. the anterior bony portion of the medial wall of the MS will be removed, .then the IT-NLD flap will be formed.The prelacrimal recess will be opened
  Interventions: Procedure: Endoscopic Approaches To Maxillary Sinus
- The canine fossa approach. (Active Comparator): It will be done either transnasally or transorally:
  ** The transoral approach through a sublabial incision : CFA consist in a trocar placed in the canine fossa.After removal of the trocar a 4-mm microdebrider blade will be placed through the passage created by the trocar.
  ** The transnasal approach: A curved incision will be made between the anterior aspect of the Inferior Turbinate and the posterior end of the nasal vestibule,the mucoperiosteum will be lifted posteriorly Then the investigators will reach the anterior wall of the maxillary sinus through bone removal which will be achieved using a gauch and hammer and a high-speed electric drill.
  Interventions: Procedure: Endoscopic Approaches To Maxillary Sinus

INTERVENTIONS:
Procedure: Endoscopic Approaches To Maxillary Sinus — The first group (group A):
  The middle meatal antrostomy approach.
  The second group (group B):
  The endoscopic prelacrimal recess approach
  The third group (group c):
  The canine fossa approach.

SUMMARY:
The aim of this study is to compare the outcomes of endoscopic pre lacrimal recess approach, canine fossa approach and middle meatal antrostomy approach regarding:

1. Assessment of the accessibility of each approach to visualize and reach the different walls and recesses of the maxillary sinus.
2. Any intraoperative or postoperative complications.
3. Any post-operative recurrence or residue detected by endoscopic examination or by MSCT scan.

DETAILED DESCRIPTION:
The maxillary sinus is the sinus most commonly affected by disease.. It varies greatly in size, shape, position and pneumatisation, not only in different individuals, but also in different sides of the same individual .

A broad spectrum of disease processes can involve the maxillary sinus, such as infective, odontogenic and neoplastic. In simple cases, a standard uncinectomy and middle meatal antrostomy may be sufficient for visualisation and clearance of disease but despite this a drawback still exists in both external and intranasal surgical procedures. Compromise of the inferior turbinate (IT) and nasolacrimal duct (NLD) is often unavoidable .

According to the anatomy of MS and the feature of diseases originated from MS assessed with multi-angulated telescopes, including 30 ,45 and 70 telescopes, with kinds of curved instruments, there are still some areas which can not be viewed and handled . Such critical areas as the inferior, lateral, anterior wall, zygomatic recess, alveolar recess and prelacrimal recess of maxillary sinus are difficult to approach. For this reason other approaches are needed like canine fossa approach (CFA), prelacrimal recess approach (PLRA) and medial maxillectomy approach.

Review of the literature revealed no meta-analysis or evidence based medicine comparing different endoscopic approaches to maxillary sinus regarding feasibility of the access to different recesses and residual lesions.

The endonasal endoscopic prelacrimal recess approach (PLRA) provides a clear view through wide access to all walls of the maxillary sinus while still preserving the nasolacrimal duct and inferior turbinate.

It enables us to accurately, mini-invade and completely remove MS lesions. It is a physiological and functional surgery, and has great advantages in treating the diseases of the nasal cavity.

Canine fossa approach (CFA) has been proposed as an alternative method of obtaining access to the maxillary antrum. Although a few studies have demonstrated the benefits of CFA in management of the severely diseased maxillary sinus, the efficacy and superiority of this method compared with conventional MMA require further investigation above all considering new microdebrider blades that can be inserted through the antrostomy.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years,
* Incidence of extensive denovo or recurrent sinonasal polyposis,
* Denovo or recurrent cases of antrochoanal polyp,
* Incidence of both denovo or recurrent allergic fungal rhinosinusitis,
* Maxillary sinus cysts and mucocoel,
* Presence of MS tumours such as inverted papilloma
* Presence of vascular tumours,
* Presence of sinonasal malignancies extending to the maxillary sinus,
* Having no contraindications for surgery under general anaesthesia.

Exclusion Criteria:

* Age less than 18 years,
* Refusal of the patient,
* Having contraindications for surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
accessibility of each endoscopic approach to visualize and reach the different walls and recesses of the maxillary sinus. | assessment will be intraoperative only during conduction of the operation.
  assessment of the accessibility and feasibility of endoscopic pre lacrimal recess approach, canine fossa approach and middle meatal antrostomy approach which will be evaluated clinically by the surgeon intraoperatively by using different types of telescopes either 0 degree telescope or multi-angulated telescopes including 30 ,45 and 70 telescopes to visualize and reach the different walls and recesses of the maxillary sinus during treatment of maxillary sinus lesions.

SECONDARY OUTCOMES:
Rate of recurrence | 6 months
  to assess the effect of each endoscopic approach on recurrence rate of maxillary sinus lesions. recurrence will be evaluated by clinical endoscopic evaluation of regular endoscopic examination first visit after one week, the second after 3 weeks and the third after 3 months. MSCT nose and paranasal sinuses will be done at the end of 6 month.

CONTACTS AND LOCATIONS:
Overall Officials: ahmed ae abdelwahab, professor, Study Chair — Assiut University
Locations (1):
- Assiut University Hospital ,Otolaryngology department., Asyut, Egypt

REFERENCES:
- [Background] Low WK. Complications of the Caldwell-Luc operation and how to avoid them. Aust N Z J Surg. 1995 Aug;65(8):582-4. doi: 10.1111/j.1445-2197.1995.tb01700.x. PMID 7661800
- [Background] Zhou B, Han DM, Cui SJ, Huang Q, Wang CS. Intranasal endoscopic prelacrimal recess approach to maxillary sinus. Chin Med J (Engl). 2013 Apr;126(7):1276-80. PMID 23557558
- [Background] Hosemann W, Scotti O, Bentzien S. Evaluation of telescopes and forceps for endoscopic transnasal surgery on the maxillary sinus. Am J Rhinol. 2003 Sep-Oct;17(5):311-6. PMID 14599136
- [Background] Anand V, Santosh S, Aishwarya A. Canine fossa approaches in endoscopic sinus surgery - our experience. Indian J Otolaryngol Head Neck Surg. 2008 Sep;60(3):214-7. doi: 10.1007/s12070-008-0080-3. Epub 2008 Oct 22. PMID 23120545
- [Background] Chen Y, Zhang H, Ge P, Wei T, Luo X, Huang P. [Combined middle meatus and expand pre-lacrimal recess-maxillary sinus approach for endoscopic maxillary sinus surgery]. Lin Chuang Er Bi Yan Hou Tou Jing Wai Ke Za Zhi. 2012 Dec;26(23):1070-2, 1076. Chinese. PMID 23451474
- [Background] Sathananthar S, Nagaonkar S, Paleri V, Le T, Robinson S, Wormald PJ. Canine fossa puncture and clearance of the maxillary sinus for the severely diseased maxillary sinus. Laryngoscope. 2005 Jun;115(6):1026-9. doi: 10.1097/01.MLG.0000162651.22019.4A. PMID 15933514